CLINICAL TRIAL: NCT03307330
Title: A Cross-sectional Study Examining Adipose Tissue in Obstructive Sleep Apnea
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Virend Somers, MD, PhD, Consultant, Professor of Medicine, Mayo Clinic
Other Study IDs: 17-003825; R01HL065176 (NIH)
Record Dates: First submitted 2017-10-06; First posted 2017-10-11 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Obstructive Sleep Apnea of Adult
Keywords: Obstructive Sleep Apnea; Adipose Tissue
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples Fat tissue Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obstructive Sleep Apnea: Obstructive sleep apnea is defined as having Apnea hypopnea index (AHI) >=5
- Non-Obstructive Sleep Apnea: Non-Obstructive sleep apnea is defined as having Apnea hypopnea index (AHI) < 5

SUMMARY:
Studies show that sleep apnea increases the risk of cardiovascular disease and is associated with obesity. However, it is unclear how sleep apnea affects fat tissue. Studies have shown that fat tissue is likely involved in developing cardiovascular disease. The purpose of this study is to see how sleep apnea changes fat tissue.

DETAILED DESCRIPTION:
In recent years, the contribution of adipose tissue to obesity-related insulin resistance (IR), diabetes mellitus and cardiovascular disease (CVD) has become clear.In particular, accumulation of damaged cells in obese and aging adipose tissue has been shown to impair adipose tissue function and may thus increase CVD risk. Cellular and molecular alterations in adipose tissue are known to contribute to adipose tissue and systemic insulin resistance, chronic inflammation, and may lead to higher blood pressure. Importantly, any clinical consequences of adipose tissue dysfunction would be compounded by the large amount, and central metabolic role, of adipose tissue in humans. However, there is a gap in our understanding of the OSA-induced changes in the adipose tissue and its implication for development of cardiometabolic disorders.

The aim of this study is to examine the cellular and molecular composition of adipose tissue in obstructive sleep apnea (OSA) subjects in comparison to adipose tissue from healthy individuals. We hypothesize that adipose tissue from OSA subjects will have a higher accumulation of markers of cellular damage with positive p16 and γH2AX. These studies will provide pivotal insights into pathways that may be targeted to reduce cardiometabolic burden in OSA population.

ELIGIBILITY:
Inclusion Criteria

* BMI ≤40 kg/m2
* Not a current smoker or tobacco user
* Individuals with treated hypertension, prehypertension, and dyslipidemia will be allowed to participate in the study
* On no prescription medications other than those medications used to treat asthma, seasonal or environmental allergies (such as Cetirizine, Fexofenadine, Desloratadine, Loratadine, etc), depression, acid reflux (such as antacids or proton pump inhibitors), topical skin treatment medications or shampoos, contraceptive pills, or intrauterine devices. Other medications may be allowed at the discretion of the study staff.
* Not pregnant or breast feeding and not intending to become pregnant or breast feed
* Ability to provide written informed consent
* If a subject is on aspirin or any other anti-inflammatory medication but free of known vascular disease and depending on the indication, the study doctor may ask the subject to suspend aspirin or anti-inflammatory therapy for 7 days prior to participation in the study. In the event that the subject does not stop the aspirin or other anti-inflammatory medication, they will not be able to participate in the study because of the risk of bleeding during the fat biopsy.

Exclusion Criteria

* Vulnerable study population will be excluded
* Presence of chronic kidney disease (creatinine >2.5 mg/dL) and/or active cancers
* Pregnancy
* Anemic (hemoglobin <12 g/dL for men and <11 g/dL for women)
* Smoking
* Use of chronic medications (statins, anti-inflammatory drugs, angiotensin II receptor blockers (ARBs) and/or angiotensin-converting enzyme (ACE) inhibitors)
* Blood or plasma donation during the past 2 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects with obstructive sleep apnea and healthy subjects without chronic diseases and interested in participating will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-01-08 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of dual positive p16^IND4A and gamma H2AX cells in adipose tissue | Day 2
  Positivity for both (p16^IND4A and γH2AX) serves as a marker of cellular damage. A fat biopsy from the abdomen and thigh will be performed to obtain up to 1 gm of adipose tissue from each site. These fat samples will be batched for analysis.

SECONDARY OUTCOMES:
Prevalence of phosphorylated p53 (pp53) in adipose tissue | Day 2
  Presence of pp53 as a ratio of phospho to total p53 to access cellular damage in adipose tissue.
24- h mean arterial pressure | Day 2
  ambulatory measure of blood pressure in mmHg
Vascular endothelial function | Day 2
  Change in Brachial artery diameter in response to hyperemia
Insulin sensitivity | Day 2
  Oral glucose tolerance testing
Body composition | Day 1
  Percentage body fat content

CONTACTS AND LOCATIONS:
Overall Officials: Virend Somers, MD., Ph.D, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States